CLINICAL TRIAL: NCT04871971
Title: Glycaemic Response and Insulinaemic Response for Nutralys S85 Plus and Whey Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Collaborators: Roquette Freres (Industry)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Principal Investigator, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CPS-20-255; WT762123 (Other: Oxford Brookes University)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — Pea Proteins; Whey; Glucose

STUDY DESIGN:
Intervention Model Description: single-blind, randomised, repeat measure, crossover design trial
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Glucose (Placebo Comparator): Glucose 50 g available carbohydrate
  Interventions: Dietary Supplement: 50 g Glucose
- 10 g NUTRALYS®S85 Plus pea protein (Experimental): 50 g available carbohydrate Glucose + 10 g NUTRALYS®S85 Plus pea protein
  Interventions: Dietary Supplement: 10 g NUTRALYS®S85 Plus pea protein
- 20 g NUTRALYS®S85 Plus pea protein (Experimental): 50 g available carbohydrate Glucose + 20 g NUTRALYS®S85 Plus pea protein
  Interventions: Dietary Supplement: 20 g NUTRALYS®S85 Plus pea protein
- 10 g Whey protein concentrate (Experimental): 50 g available carbohydrate Glucose + 10 g Whey protein concentrate
  Interventions: Dietary Supplement: 10 g Whey protein concentrate
- 20 g Whey protein concentrate (Experimental): 50 g available carbohydrate Glucose + 20 g Whey protein concentrate
  Interventions: Dietary Supplement: 20 g Whey protein concentrate

INTERVENTIONS:
Dietary Supplement: 10 g NUTRALYS®S85 Plus pea protein — To determine the glycaemic response and insulinaemic response to 50g Glucose + 10 g NUTRALYS®S85 Plus pea protein.
  Arms: 10 g NUTRALYS®S85 Plus pea protein
Dietary Supplement: 20 g NUTRALYS®S85 Plus pea protein — To determine the glycaemic response and insulinaemic response to 50g Glucose + 20 g NUTRALYS®S85 Plus pea protein.
  Arms: 20 g NUTRALYS®S85 Plus pea protein
Dietary Supplement: 10 g Whey protein concentrate — To determine the glycaemic response and insulinaemic response to 50g Glucose + 10 g Whey protein concentrate.
  Arms: 10 g Whey protein concentrate
Dietary Supplement: 20 g Whey protein concentrate — To determine the glycaemic response and insulinaemic response to 50g Glucose + 20 g Whey protein concentrate.
  Arms: 20 g Whey protein concentrate
Dietary Supplement: 50 g Glucose — To determine the glycaemic response and insulinaemic response to 50g Glucose
  Arms: Glucose

SUMMARY:
A comparison of the glycaemic response and insulinaemic response to glucose, Nutralys S85 Plus pea protein and whey protein using a single-blind, randomised, repeat measure, crossover design trial.

DETAILED DESCRIPTION:
A single-blind, randomised, repeat measure, crossover design trial will be used to study the glycaemic response and insulinaemic response following consumption of five products: one reference product (50 g available carbohydrate Glucose) and four test products (50 g available carbohydrate Glucose with 10 g NUTRALYS®S85 Plus pea protein, 50 g available carbohydrate Glucose with 20 g NUTRALYS®S85 Plus pea protein, 50 g available carbohydrate Glucose with 10 g Whey protein concentrate and 50 g available carbohydrate Glucose with 20 g Whey protein concentrate).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years
* Body mass index (BMI) less than 30kg/m2

Exclusion Criteria:

* Pregnant or lactating
* Fasting blood glucose value > 6.1 mmol/l
* Any known food allergy or intolerance
* Medical condition(s) or medication(s) known to affect glucose regulation or appetite and/or which influence digestion and absorption of nutrients
* Known history of diabetes mellitus or the use of antihyperglycaemic drugs or insulin to treat diabetes and related conditions
* Major medical or surgical event requiring hospitalization within the preceding 3 months
* Use of steroids, protease inhibitors or antipsychotics (all of which have major effects on glucose metabolism and body fat distribution)
* Unable to comply with experimental procedures or did not follow GR testing safety guidelines.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose response from baseline for 3 hours | 3 hours
  Change in postprandial blood glucose response from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Change in plasma insulin response from baseline for 3 hours | 3 hours
  Change in postprandial plasma insulin response from baseline was measured at 15 min, 30 min, 45 min, 1 hour, 1.5 hours, 2 hours, 2.5 hours and 3 hours
Area under the blood glucose concentration versus time curve | 3 hours
  Area under the blood glucose concentration versus time curve was calculated by trapezoidal rule
Area under the plasma insulin concentration versus time curve | 3 hours
  Area under the plasma insulin concentration versus time curve was calculated by trapezoidal rule
Peak blood glucose concentration (Cmax) | 0-3 hours
  Peak blood glucose concentration (Cmax) after consumption of the test food
Peak plasma insulin concentration (Cmax) | 0-3 hours
  Peak plasma insulin concentration (Cmax) after consumption of the test food
Time of blood glucose peak (Tmax) | 0-3 hours
  Time of blood glucose peak after consumption of the test food
Time of plasma insulin peak (Tmax) | 0-3 hours
  Time of plasma insulin peak after consumption of the test food

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Thondre, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siahanidou T, Margeli A, Kappis A, Papassotiriou I, Mandyla H. Circulating visfatin levels in healthy preterm infants are independently associated with high-density lipoprotein cholesterol levels and dietary long-chain polyunsaturated fatty acids. Metabolism. 2011 Mar;60(3):389-93. doi: 10.1016/j.metabol.2010.03.002. Epub 2010 Mar 31. PMID 20359723
- See also: Food Products-Determination of the glycaemic index (GI) and recommendation for food classification. — http://www.iso.org/standard/43633.html

DOCUMENTS (1):
  • Informed Consent Form (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT04871971/ICF_000.pdf